CLINICAL TRIAL: NCT00457509
Title: Safety and Immunogenicity of H5N1 Adjuvanted, Inactivated, Split-Virion Pandemic Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GPF01
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Pandemic Influenza; Influenza A Virus Infection; Orthomyxoviridae Infections
Keywords: Pandemic influenza; Avian influenza; Orthomyxoviridae Infections; A/H5N1
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza in Birds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Dose 1 with Adjuvant
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant
- Group 2 (Experimental): Dose 2 with adjuvant
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant
- Group 3 (Experimental): Dose 3 with adjuvant
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant
- Group 4 (Experimental): Dose 4 with adjuvant
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant
- Group 5 (Active Comparator): Control
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza vaccine

INTERVENTIONS:
Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant — 0.5 mL, Intramuscular
  Arms: Group 1
Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant — 0.5 mL, Intramuscular
  Arms: Group 2
Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant — 0.5 mL, Intramuscular
  Arms: Group 3
Biological: A/H5N1 inactivated, split-virion influenza vaccine+Adjuvant — 0.5 mL, Intramuscular
  Arms: Group 4
Biological: A/H5N1 inactivated, split-virion influenza vaccine — 0.5 mL, Intramuscular
  Arms: Group 5

SUMMARY:
The purpose of this study is to test different adjuvanted vaccine formulations as a two-dose schedule in immunologically naïve adults against one vaccine formulation without adjuvant in terms of tolerance and immunogenicity

Primary Objective:

To describe the safety profile and immunogenicity following each injection.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 40 years on day of inclusion
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative urine pregnancy test.

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Previous participation in a clinical trial involving an investigational flu pandemic vaccine.
* Vaccination with an influenza vaccine during the past 6 months
* Any vaccination in the 4 weeks preceding the first trial vaccination
* Vaccination planned in the 4 weeks following any trial vaccination
* Breast-feeding.
* For a woman of child-bearing potential, the absence of an effective method of contraception or abstinence non observed for at least 4 weeks prior to the first vaccination and at least 4 weeks after the last vaccination.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy.
* Known human immunodeficiency virus (HIV), hepatitis B (AgHBs) or hepatitis C seropositivity.
* Known systemic hypersensitivity to egg proteins, chick proteins, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Blood or blood-derived products received in the past 3 months.
* Febrile illness (temperature ≥ 37.5°C) on the day of inclusion.
* Laboratory abnormalities considered clinically significant upon the Investigator's judgment in blood sample taken at screening (for Step 1 only)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2007-01; Primary Completion 2009-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety of A/H5N1 Inactivated split influenza virus vaccine | Entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (3):
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven

REFERENCES:
- [Derived] Levie K, Leroux-Roels I, Hoppenbrouwers K, Kervyn AD, Vandermeulen C, Forgus S, Leroux-Roels G, Pichon S, Kusters I. An adjuvanted, low-dose, pandemic influenza A (H5N1) vaccine candidate is safe, immunogenic, and induces cross-reactive immune responses in healthy adults. J Infect Dis. 2008 Sep 1;198(5):642-9. doi: 10.1086/590913. PMID 18576945
- See also: Related Info — http://www.sanofipasteur.com